CLINICAL TRIAL: NCT04380987
Title: Luxembourg Cohort of Positive Patients for COVID-19: a Stratification Study to Predict Patient Prognosis
Acronym: Predi-COVID
Status: Completed | Type: Observational
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Centre Hospitalier du Luxembourg (Other); Hopitaux Robert Schuman (Luxembourg) (Unknown); Laboratoire National de Santé (Luxembourg) (Unknown); University of Luxembourg (Other)
Responsible Party: Sponsor
Other Study IDs: Predi-Covid
Record Dates: First submitted 2020-04-30; First posted 2020-05-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Covid19
Keywords: Severity factors; Patient stratification; Digital
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological/Vaccine: Biological sampling For every symptomatic adult tested positive by RTqPCR, up to 45 mL of blood will be taken, nasopharyngeal and oropharyngeal swab will be performed, an induced sputum and a stool samples will be recovered at the inclusion. As follow-up, 3 weeks after inclusion, up to 45 mL of blood will be taken and a new induced sputum will be recovered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Predicovid
  Interventions: Biological: Biological sampling

INTERVENTIONS:
Biological: Biological sampling — For every symptomatic adult tested positive by RTqPCR, up to 45 mL of blood will be taken, nasopharyngeal and oropharyngeal swab will be performed, an induced sputum and a stool samples will be recovered at the inclusion. As follow-up, 3 weeks after inclusion, up to 45 mL of blood will be taken and a new induced sputum will be recovered.

SUMMARY:
Predi-COVID is a prospective cohort study composed of people positively tested for COVID-19 in Luxembourg, followed digitally for monitoring participants' health evolution and symptoms at home. Participants will be actively followed for 14 days from the time of confirmation of diagnosis, whether they are at the hospital or at home in isolation or quarantine. Short evaluations will be also performed at week 3 and week 4 and then monthly for a period up to 12 months to assess potential long term consequences of COVID-19. A subsample of 200 participants will be contacted to integrate complementary clinical data and collect samples.

The study aims at identifying factors associated with the COVID-19 disease severity. COVID-19 patients with severity criteria will be compared to patients with mild disease managed at home.

A deep phenotyping related to the symptoms of the disease as well as biosampling allowing for laboratory-based and computational analytics will be performed.

DETAILED DESCRIPTION:
The objective is to recruit virtually all COVID-19 positive persons in Luxembourg.

The sub-sample of a minimum of 200 COVID-19 positive persons in Predi-COVID study would allow to find a risk ratio of severe disease above 2 for the selected risk factor with a power of 80% when the prevalence of the disease is above 7%.

For every symptomatic adult tested positive by RTqPCR, biological samples will be collected at the inclusion and as follow-up 3 weeks after inclusion.

For patients at home, an experienced nurse from CIEC will perform the sampling, using all the required precautions and protections in the actual context.

For hospitalised patients, a simplified sampling strategy will be put in place and adapted to the patient state, the workload of staff and adapted constantly depending on the evolution of the epidemy.

Data will be collected through 3 different ways :

1. Questionnaires : health status monitoring data with daily questionnaires during the 14 first days following diagnosis, weekly questionnaires at week 3 and 4 and monthly questionnaires from month 2 to month 12.
2. Adapted ISARIC eCRF for patients at hospital (during all hospital stay) and at inclusion for patients included from home.
3. Smartphone application (LIH in-house solution) : innovative data (voice recordings, geolocation and mini-questionnaires).

An ancillary study will be added (Predi-COVID-H):

Predi-COVID-H is an ancillary cohort study composed of Household members of index cases to monitor symptoms and disease outbreak in this high-risk population. For every asymptomatic member of the family of a "case" included in the Predi-COVID sub-sample (a "contact"), clinical as well as socio-economic characteristics will be collected. Biological samples will also be collected at the same time as the "case" visit by nurses and up to 30 ml of blood will be taken at baseline, for serology. IgG and/or IgA seropositive "contacts" will be proposed to be enrolled in the Predi-COVID study. For IgG and IgA seronegative "contacts", a second serology will be planned 2 weeks later, up to 30 mL of blood will be collected. If they become IgG and/or IgA seropositive, they will be proposed to be enrolled in the Predi-COVID study. IgG and IgA seronegative "contacts" will be followed digitally

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection as determined by PCR, performed by one of the certified laboratories in Luxembourg
* Signed informed consent form
* Age ≥18 years old
* Hospitalized or at home

Exclusion Criteria:

* Patients not understanding French or German
* Patients already included in an interventional study on Covid-19 (Discovery or other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years old) patients with confirmed SARS-CoV-2 infection, hospitalized or at home.
Sampling Method: Non-Probability Sample
Enrollment: 1366 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Description of clinical manifestations | 1 year
  Number of symptoms associated with Covid-19

SECONDARY OUTCOMES:
Clinical aggravation of the infection | 1 year
  Number of hospitalizations
Discharge of hospitalization | 1 year
  Number of discharges
Death | 1 year
  Number of deaths
Description of biological manifestations | 1 year
  Whole blood count parameters
Description of biological manifestations | 1 year
  Plasma cytokine levels
Description of biological manifestations | 1 year
  Antibodies to SARS-Cov2
Patient-related prognostic factors | 1 year
  HLA genotypes
Patient-related prognostic factors | 1 year
  Coinfections
Virus-related prognostic factors | 1 year
  Virus mutations
Vocal biomarker of Covid-19 related respiratory complications | 1 year
  Audio feature extracted from 30 seconds recordings of participants' voice reading a prespecified text, collected throughout the CoLIVE LIH smartphone app.

CONTACTS AND LOCATIONS:
Locations (1):
- Luxembourg Institute of Health, Luxembourg, Luxembourg

REFERENCES:
- [Derived] Fischer A, Zhang L, Elbeji A, Wilmes P, Snoeck CJ, Larche J, Oustric P, Ollert M, Fagherazzi G. Trajectories of persisting Covid- 19 symptoms up to 24 months after acute infection: findings from the Predi-Covid cohort study. BMC Infect Dis. 2025 Apr 25;25(1):603. doi: 10.1186/s12879-025-11023-0. PMID 40281467
- [Derived] Elbeji A, Zhang L, Higa E, Fischer A, Despotovic V, Nazarov PV, Aguayo G, Fagherazzi G. Vocal biomarker predicts fatigue in people with COVID-19: results from the prospective Predi-COVID cohort study. BMJ Open. 2022 Nov 22;12(11):e062463. doi: 10.1136/bmjopen-2022-062463. PMID 36414294
- [Derived] Higa E, Elbeji A, Zhang L, Fischer A, Aguayo GA, Nazarov PV, Fagherazzi G. Discovery and Analytical Validation of a Vocal Biomarker to Monitor Anosmia and Ageusia in Patients With COVID-19: Cross-sectional Study. JMIR Med Inform. 2022 Nov 8;10(11):e35622. doi: 10.2196/35622. PMID 36265042
- [Derived] Fischer A, Zhang L, Elbeji A, Wilmes P, Oustric P, Staub T, Nazarov PV, Ollert M, Fagherazzi G. Long COVID Symptomatology After 12 Months and Its Impact on Quality of Life According to Initial Coronavirus Disease 2019 Disease Severity. Open Forum Infect Dis. 2022 Aug 5;9(8):ofac397. doi: 10.1093/ofid/ofac397. eCollection 2022 Aug. PMID 35983269
- [Derived] Malisoux L, Backes A, Fischer A, Aguayo G, Ollert M, Fagherazzi G. Associations between physical activity prior to infection and COVID-19 disease severity and symptoms: results from the prospective Predi-COVID cohort study. BMJ Open. 2022 Apr 29;12(4):e057863. doi: 10.1136/bmjopen-2021-057863. PMID 35487745
- [Derived] Fagherazzi G, Fischer A, Betsou F, Vaillant M, Ernens I, Masi S, Mossong J, Staub T, Brault D, Bahlawane C, Rashid MA, Ollert M, Gantenbein M, Huiart L. Protocol for a prospective, longitudinal cohort of people with COVID-19 and their household members to study factors associated with disease severity: the Predi-COVID study. BMJ Open. 2020 Nov 23;10(11):e041834. doi: 10.1136/bmjopen-2020-041834. PMID 33234656